CLINICAL TRIAL: NCT01975909
Title: Transcranial Magnetic Stimulation (TMS) in Spino-Cerebellar Ataxia
Brief Title: Transcranial Magnetic Stimulation in Spino-Cerebellar Ataxia
Acronym: TMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Alvaro Pascual-Leone, Professor of Neurology, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2013P000233; 1R21NS085491-01 (NIH)
Record Dates: First submitted 2013-09-24; First posted 2013-11-05 (Estimated); Results first posted 2017-05-30 (Actual); Last update posted 2017-05-30 (Actual); Status verified 2017-04

CONDITIONS: Spinocerebellar Ataxia
Keywords: Spinocerebellar Ataxia; SCA; Ataxia; Transcranial Magnetic Stimulation; TMS
MeSH Terms: conditions — Spinocerebellar Ataxias; Ataxia | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Transcranial Magnetic Stimulation (TMS) (Active Comparator): A Magstim 200 (Magstim, UK) and 14cm circular coil positioned tangential to the head will be used to deliver stimuli at 100% of maximum stimulator output. Transcranial Magnetic Stimulation will be applied to three regions: 1) 4cm lateral to the right of the inion, 2) centered on the inion, 3) 4cm lateral to the left of the inion. Five pulses separated by 6 seconds will be delivered with a counter-clockwise current, followed by the same five pulses delivered with a clockwise current, for a total of 10 pulses per region, and 30 pulses per session.
  Interventions: Device: Transcranial Magnetic Stimulation
- Sham Transcranial Magnetic Stimulation (Sham Comparator): A sham condition of Transcranial Magnetic Stimulation will be used and follow the same protocol as the active stimulation; however no magnetic pulses will be delivered through the scalp.
  Interventions: Device: Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation — 0.2 Hz (5 pulses every six seconds in a counter-clockwise current, followed by the same five pulses in a clockwise current); 10 pulses per region, 30 pulses per session; 5 days a week for 4 weeks.
  Other Names: Magstim 200

SUMMARY:
Spinocerebellar Ataxia (SCA) refers to a family of genetic diseases that cause progressive problems with gait and balance, as well as other debilitating symptoms. This is a randomized controlled pilot study to test a novel therapeutic intervention that uses noninvasive magnetic brain stimulation to improve functional outcomes in patients with SCA. The study will include quantitative evaluations of gait, balance, and brain physiology to examine possible objective end-points for a future, larger multi-site clinical trial. The investigators anticipate that patients receiving the real intervention will show a functional gain.

DETAILED DESCRIPTION:
Spinocerebellar Ataxia (SCA) refers to a family of genetic diseases that cause progressive problems with gait and balance, as well as other debilitating symptoms. There is no cure for SCA and a lack of an effective symptomatic treatment.

Investigators will recruit 20 patients with genetically-confirmed SCA to use a novel approach - noninvasive transcranial magnetic stimulation (TMS) - to improve balance, gait, and posture in patients with SCA. Half will be randomly assigned to a real intervention, and half to a sham (control) intervention. The TMS intervention will consist of 20 stimulation sessions over a four week period. At baseline and follow-up, patients will undergo comprehensive assessments including several SCA rating scales, along with sophisticated tests of balance (ie. walking, standing, and muscle coordination). Patients will also complete a series of neurophysiologic tests to evaluate the function of the cerebellum and its connections before and after the intervention.

Investigators anticipate patients receiving real TMS will show better balance, fewer falls, and improved mobility, while those undergoing sham stimulation will show no benefits. If our prediction is correct, this study will provide evidence-based support for a new treatment to improve the lives of patients with SCA.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients with ataxia as diagnosed by a movement disorder specialist and confirmed by clinically obtained genetic testing of the patient and/or in a first-degree relative of the patient.
* Women of child-bearing potential must use a reliable method of contraception and must provide a negative pregnancy test at entry into the study
* Stable on doses of all medications for at least 30 days prior to study entry and for the duration of the study
* The ability to ambulate
* A score of three or higher (worse) on the 'gait' subsection of the Scale of the Assessment and Rating of Ataxia (SARA) rating scale.

Exclusion Criteria:

* Any unstable illness or concomitant medical condition that, in the investigator's opinion, precludes participation in this study, including disorders that may affect gait or balance (i.e., stroke, arthritis, etc).
* The presence of clinically significant abnormalities on screening CBC, CMP or EKG.
* Pregnancy or lactation
* Concurrent participation in another clinical study
* A history of substance abuse
* The presence of psychosis, bipolar disorder, untreated depression (BDI greater than or equal to 21), or history of suicide attempt.
* Dementia or other psychiatric illness that prevents the patient from giving informed consent (Mini Mental Status Exam score less than 24).
* Legal incapacity or limited legal capacity.
* Ataxia derived from any cause other than genetically-confirmed SCA (including but not limited to alcoholism, head injury, Multiple Sclerosis, olivo-ponto-cerebellar atrophy or multiple system atrophy).
* No medication is an absolute exclusion from TMS. Medications will be reviewed by the responsible MD and a decision about inclusion will be made based on the following:

  1. The patient's past medical history, drug dose, history of recent medication changes or duration of treatment, and combination with other CNS active drugs.
  2. The published TMS guidelines review of medications to be considered with TMS.
* History of seizures, diagnosis of epilepsy, history of abnormal (epileptiform) EEG.
* TMS and MRI-Specific exclusion criteria including:

  1. Known metal in the head (such as a surgical aneurysm clip) or a history of prior neurosurgical procedures.
  2. Ferromagnetic bioimplants activated by any electronic, mechanical or magnetic means, such as cochlear implants, pacemakers, medication pumps, vagal stimulators, deep brain stimulators, neurostimulators, biostimulators, or ventriculo-peritoneal shunts.
  3. Subjects who have or might have bullet fragments or other shrapnel (veterans or workers exposed to metal in their work environment).
  4. Subjects with metallic paint (e.g. color contact lenses, tattoos, metallic eyeliner)
  5. Subjects expressing significant claustrophobia.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-09; Primary Completion 2016-10 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alvaro Pascual-Leone, MD, PhD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Manor B, Greenstein PE, Davila-Perez P, Wakefield S, Zhou J, Pascual-Leone A. Repetitive Transcranial Magnetic Stimulation in Spinocerebellar Ataxia: A Pilot Randomized Controlled Trial. Front Neurol. 2019 Feb 12;10:73. doi: 10.3389/fneur.2019.00073. eCollection 2019. PMID 30809184
- See also: Information on TMS and the lab conducting the study — http://tmslab.org/
- See also: Information on Ataxia — http://www.ataxia.org/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Transcranial Magnetic Stimulation (TMS) | Sham Transcranial Magnetic Stimulation
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Transcranial Magnetic Stimulation (TMS) | Sham Transcranial Magnetic Stimulation | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.3 (10.1) | 48.6 (4.8) | 50.6 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 16
  Male | 2 | 2 | 4
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline to Post Treatment on the Scale for the Assessment and Rating of Ataxia (SARA)
Description: Assess 8 items: gait, stance, sitting, speech, dysmetria, kinetic tremor, pro- and supinations of the hand, and the heel-shin slide. Each item is scored by the physician on a 4 to 8 numerical scale based upon the amount of dysfunction observed while performing the task. The maximum possible score for the total scale is 40. Lower scores of SARA represents better task performance.
Time Frame: Baseline and 1 week post treatment
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Transcranial Magnetic Stimulation (TMS) | Sham Transcranial Magnetic Stimulation
Number analyzed (Participants) | 10 | 10
percentage change | -25.9 (16.4) | -27.8 (9.0)
Statistical Analysis 1: Comparison: Transcranial Magnetic Stimulation (TMS) vs Sham Transcranial Magnetic Stimulation; Test type: Equivalence — We hypothesized that the real TMS would improve the performance of SARA (i.e., greater percent decrease of SARA score from baseline) as compared to the sham TMS; p = 0.29, t-test, 2 sided

2. Secondary Outcome: Percent Change From Baseline to Post Treatment on the Timed 25-Foot Walk
Description: A quantitative assessment of mobility and leg function. Two trials of patients walking along a 25ft course as quickly and safely as possible. Time taken to complete course will be recorded and averaged across trials.
Time Frame: Baseline and 1 week post treatment
Measure: Mean (Standard Deviation); unit: percentage change of maximum gait speed
Arm/Group | Transcranial Magnetic Stimulation (TMS) | Sham Transcranial Magnetic Stimulation
Number analyzed (Participants) | 10 | 10
percentage change of maximum gait speed | 7.8 (12.0) | 2.2 (25.6)
Statistical Analysis 1: Comparison: Transcranial Magnetic Stimulation (TMS) vs Sham Transcranial Magnetic Stimulation; Test type: Equivalence — We hypothesized that the real TMS would improve the performance of 25-foot walking test (i.e., greater percent increase of walking speed from baseline) as compared to the sham TMS; p = 0.47, t-test, 2 sided

3. Secondary Outcome: Percent Change From Baseline to Post Treatment on the 9-hole Peg Test
Description: The test consists of a block with nine holes, into which the subject places and then removes 9 pegs. The time taken to complete the test will be recorded.
Time Frame: Baseline and 1 week post treatment
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Transcranial Magnetic Stimulation (TMS) | Sham Transcranial Magnetic Stimulation
Number analyzed (Participants) | 10 | 10
percentage change | 0.7 (5.1) | -6.7 (7.2)
Statistical Analysis 1: Comparison: Transcranial Magnetic Stimulation (TMS) vs Sham Transcranial Magnetic Stimulation; Test type: Equivalence — We hypothesized that the real TMS would improve the performance of 9-hole peg test (i.e., greater percent decrease of time to complete the test from baseline) as compared to the sham TMS; p = 0.12, t-test, 2 sided

4. Other Pre Specified Outcome: Percent Change From Baseline to Post Treatment on Gait Speed in 90 Second Walking Test
Description: Two 90 second trials of walking at a preferred speed along a 80x4m indoor hallway. A wireless Noraxon DTS system (Noraxon Inc, Scottsdale, AZ) will be used simultaneously and continuously record bilateral foot placements, 3-dimensional trunk accelerations, and lower-extremity surface electromyography of eight muscles.
Time Frame: Baseline and 1 week post treatment
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Transcranial Magnetic Stimulation (TMS) | Sham Transcranial Magnetic Stimulation
Number analyzed (Participants) | 10 | 10
percentage change | 4.2 (17.9) | 5.3 (13.1)
Statistical Analysis 1: Comparison: Transcranial Magnetic Stimulation (TMS) vs Sham Transcranial Magnetic Stimulation; Test type: Equivalence — We hypothesized that the real TMS would improve the performance of 90-second walking test (i.e., greater percent increase of walking speed from baseline) as compared to the sham TMS; p = 0.69, t-test, 2 sided

5. Other Pre Specified Outcome: Percent Change From Baseline to Post Treatment on Standing Postural Control
Description: Postural control - assessed by measuring standing postural sway (ie., center-of pressure fluctuations) during two, 30second trials of standing with eyes open on a stationary force platform (AMTI, Watertown, MA).
Time Frame: Baseline and 1 week post treatment
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Transcranial Magnetic Stimulation (TMS) | Sham Transcranial Magnetic Stimulation
Number analyzed (Participants) | 10 | 10
percentage change | -21.5 (14.9) | 13.2 (29.7)
Statistical Analysis 1: Comparison: Transcranial Magnetic Stimulation (TMS) vs Sham Transcranial Magnetic Stimulation; Test type: Equivalence — We hypothesized that the real TMS would improve the standing postural control stability (i.e., greater percent decrease increase of postural sway speed from baseline) as compared to the sham TMS; p = 0.009, t-test, 2 sided

6. Other Pre Specified Outcome: Percent Change From Baseline to Post Treatment on Mobility and Turning
Description: Mobility and turning is assessed by the timed up-and-go test (Podsiadlo & Richardson, 1991). The participant will be seated in an armed chair. On the word "go," the subject will stand up using the arm rests if needed, walk (with assistive device if needed) around a cone placed three meters in front of the chair, return and sit down as quickly as possible.
Time Frame: Baseline and 1 week post treatment
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Transcranial Magnetic Stimulation (TMS) | Sham Transcranial Magnetic Stimulation
Number analyzed (Participants) | 10 | 10
percentage change | -12.8 (11.7) | -9.3 (15.5)
Statistical Analysis 1: Comparison: Transcranial Magnetic Stimulation (TMS) vs Sham Transcranial Magnetic Stimulation; Test type: Equivalence — We hypothesized that the real TMS would improve the performance of TUG test (i.e., greater percent decrease of time to complete TUG test from baseline) as compared to the sham TMS; p = 0.18, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 2 months
Arm/Group | Transcranial Magnetic Stimulation (TMS) | Sham Transcranial Magnetic Stimulation
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No